CLINICAL TRIAL: NCT00445497
Title: A Prospective Randomised Phase III Trial of Early Hospital Discharge Versus Standard Inpatient Management of Cancer Patients With Low-Risk Febrile Neutropenia Receiving Oral Antibiotics. Oral Antibiotics for Neutropenic Sepsis Giving Early Hospital Discharge [ORANGE]
Brief Title: Early Hospital Discharge or Standard Inpatient Care in Cancer Patients Receiving Antibiotics for Febrile Neutropenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clatterbridge Centre for Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CRUK-MX3006; CDR0000533828 (Registry Identifier: PDQ (Physician Data Query)); CRUK-ORANGE; ISRCTN18467252; EU-20707
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-05

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Neutropenia; Psychosocial Effects of Cancer and Its Treatment; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; intraocular lymphoma; nodal marginal zone B-cell lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; small intestine lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV small lymphocytic lymphoma; Waldenström macroglobulinemia; unspecified adult solid tumor, protocol specific; neutropenia; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Hodgkin lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage II adult Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neutropenia; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell | interventions — Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin; Psychiatric Rehabilitation

INTERVENTIONS:
Drug: amoxicillin-clavulanate potassium
Drug: ciprofloxacin
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Finishing an antibiotic regimen at home may be as effective as receiving it in the hospital. It is not yet known whether early hospital discharge is as effective as standard inpatient care in cancer patients receiving antibiotics for febrile neutropenia.

PURPOSE: This randomized phase III trial is studying early hospital discharge and comparing it with standard inpatient care in cancer patients receiving antibiotics for febrile neutropenia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify cancer patients who are low-risk inpatients and meet criteria for early discharge (i.e., symptomatic improvement and temperature ≤ 37.8°C) after receiving oral antibiotics for febrile neutropenia.

OUTLINE: This is a randomized, prospective, multicenter study. Patients are stratified by disease type (lymphoma vs solid tumor), duration of registration (< 48 hours vs > 48 hours), and participating center.

Patients receive oral amoxicillin-clavulanate potassium 3 times daily and oral ciprofloxacin twice daily on admission to the hospital. Treatment continues for 7 days in the absence of clinical deterioration or unacceptable toxicity. Patients are assessed as inpatients after ≥ 24 and up to 72 hours after the first antibiotic dose. Patients showing clear response (i.e., symptomatic improvement irrespective of neutrophil recovery, temperature ≤ 37.8 C for 24 hours) and who continue to meet study eligibility criteria are randomized to 1 of 2 arms.

* Arm I (early discharge): Patients are discharged home and instructed to remain in daily contact with hospital staff to report temperature and symptoms until completion of oral antibiotic regimen.
* Arm II (standard management): Patients continue their antibiotic course in hospital and are discharged according to local guidelines and the following additional criteria: subjective improvement, afebrile (≤ 37°C for 24 hours), and absolute neutrophil count ≥ 500/mm³ and rising.

Patients in both arms complete a daily diary documenting daily temperature readings, symptoms, and toxicities. Patients also complete a Health Questionnaire and a Cancer Worries Inventory Booklet at baseline, in the hospital immediately after randomization, and at completion of oral antibiotics or resolution of neutropenic febrile episode.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor or lymphoma AND meets the following criteria:

  * Low-risk patient, defined as Multinational Association for Supportive Care in Cancer prognostic index score ≥ 21
  * Presents with neutropenic fever defined as follows:

    * Absolute neutrophil count ≤ 500/mm³ OR < 1,000/mm³ but anticipated to fall to ≤ 500/mm³ within 24 hours of study entry
    * Temperature ≥ 38.5°C on a single measurement or ≥ 38.0°C on > 1 occasion (one of which could be measured by the patient prior to admission) ≥ 1 hour apart
  * Undergoing concurrent cytotoxic chemotherapy for treatment of solid tumors or lymphoma
* No leukemia

PATIENT CHARACTERISTICS:

* Compliant and appropriate for early discharge
* Able to read a thermometer (patient or caregiver)
* Able to tolerate oral medication
* Must have a responsible adult caregiver if eligible for early discharge
* No known allergy to oral antibiotics or penicillin
* No requirement for IV fluid support
* No central venous catheter-associated infection or evidence of infection not amenable to treatment by study antibiotics
* No neutropenic fever at high risk of complications
* No associated comorbidity that requires hospitalization and management
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior participation in this study for neutropenic episode
* No prior bone marrow transplantation or peripheral blood stem cell transplantation
* No prior treatment for leukemia
* More than 72 hours since prior antibiotics, including prophylactic antibiotics

  * Prophylactic septrin (for pneumocystis), acyclovir, or antifungals are allowed
* No concurrent granulocyte colony-stimulating factor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Total number of days of hospitalization (including unplanned readmission) (randomized patients)
Incidence of serious adverse events (randomized and registered patients)

SECONDARY OUTCOMES:
Incidence of treatment failure as defined by the necessity for change in antibiotic therapy (randomized and registered patients)
Incidence of unplanned readmissions (randomized patients)
Patient acceptability of randomized discharge policy as measured by Health Questionnaire, Cancer Worries Inventory Booklet, and Patient Daily Diary (randomized patients)
Toxicity attributed to oral antibiotic therapy as measured by NCI CTCAE v3.0 (randomized and registered patients)
Health service costs (randomized patients)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Marshall, MD, Study Chair — Clatterbridge Centre for Oncology
Locations (10):
- United Kingdom (10):
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Leicester Royal Infirmary, Leicester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northampton General Hospital, Northampton, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Airedale General Hospital, West Yorkshire, England
  - Western Infirmary, Glasgow, Scotland
  - Ysbyty Gwynedd, Bangor, Wales